CLINICAL TRIAL: NCT00725387
Title: Combined F-18 NaF and F-18 FDG PET/CT for Evaluation of Malignancy
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: VAR0024; 98043 (Other: Stanford University Alternate IRB Approval No.); SU-07232008-1266 (Other: Stanford University)
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Fluorine-18 Fluorodeoxyglucose (F-18 FDG) PET/CT is established as a powerful imaging tool for cancer detection and monitoring response to therapy. Sodium Fluorine-18 (F-18) was used in the 1970s for bone scanning and can be used as a skeletal tracer in current PET/CT scanners. The combined administration of F-18 and F-18 FDG in a single PET/CT scan for cancer detection was not attempted to date. We hope to learn what is the best approach for detection of cancer and thus to improve cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18-year-old, diagnosed with cancer
* Patients must understand and voluntarily sign an Informed Consent form after the contents have been fully explained to them

Exclusion Criteria:

* Patients who cannot complete a PET/CT scan
* Pregnant women
* Healthy volunteers
* Patients participating in other research studies

The subjects will not be paid to participate in this protocol. No costs will be charged to the subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must be referred for evaluation of bone metastases.
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Percent of patients with evidence of new lesions on combined F-18/F-18 FDG PET/CT. | not defined

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Iagaru M.D, Principal Investigator — Stanford University
Locations (5):
- Stanford University School of Medicine, Stanford, California, United States
- Aalborg Hospital, Aalborg, Denmark
- Apollo Hospital, Chennai, India
- Coimbra University Hospital, Coimbra, Portugal
- Pretoria Academic Hospital, Pretoria, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iagaru A, Mittra E, Mosci C, Dick DW, Sathekge M, Prakash V, Iyer V, Lapa P, Isidoro J, de Lima JM, Gambhir SS. Combined 18F-fluoride and 18F-FDG PET/CT scanning for evaluation of malignancy: results of an international multicenter trial. J Nucl Med. 2013 Feb;54(2):176-83. doi: 10.2967/jnumed.112.108803. Epub 2012 Dec 14. PMID 23243299